CLINICAL TRIAL: NCT02849470
Title: Biocellular Regenerative Therapy in Hair Loss: Use of High Density Platelet-Rich Plasma Concentrates and Cell-Enriched Emulsified Adipose-Derived Tissue Stromal Vascular Fraction
Brief Title: AGA Biocellular Stem/Stromal Hair Regenerative Study
Acronym: STRAAND
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated by researchers without submission of patient admission to study. COVID complicated continuing search for qualified candidates
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Ministry of Health, Honduras (Other Government); Robert W. Alexander, MD (Unknown); Terry, Glenn C., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GARM 6.1.16
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hair Disease
Keywords: Adipose Stem/Stromal Cells; PRP; SVF; Cell Therapy; Alopecia; GF
MeSH Terms: conditions — Hair Diseases; Alopecia | interventions — Injections, Intradermal; Digestion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ARM 1 (Active Comparator): Control: 1) HD-PRP + Matristem Matrix (ACell) (Current Standard of Care); 2) Intradermal injections of hair loss 3) Platelet Rich Plasma 4) Matristem Matrix (ACell)
  Interventions: Procedure: Intradermal Injection in hair loss; Procedure: Platelet Rich Plasma; Procedure: MatriStem Matrix (ACell) - Current Standard of Care; Procedure: HD-PRP (High Density Platelet Rich Plasma)
- ARM 2 (Active Comparator): 1. Experimental: HD-PRP + Emulsified AD-tSVF;
     Intervention:
  2. Platelet Rich Plasma
  3. Adipose Derived Stem/Stromal Cells
  4. Intradermal injections of hair loss
  Interventions: Procedure: Intradermal Injection in hair loss; Procedure: Platelet Rich Plasma; Procedure: Adipose Derived Stem/Stromal Cells; Procedure: HD-PRP (High Density Platelet Rich Plasma); Procedure: Emulsified AD-tSVF
- ARM 3 (Experimental): Experimental: HD- PRP + Emulsified AD-tSVF + Emulsified AD-cSVF; Intervention: Intradermal injections of hair loss
  1. Platelet Rich Plasma
  2. Adipose Derived Stem/Stromal Cells
  3. Stem/Stromal Cell Isolation
  4. Intradermal injections of hair loss
  Interventions: Procedure: Intradermal Injection in hair loss; Procedure: Platelet Rich Plasma; Procedure: Adipose Derived Stem/Stromal Cells; Procedure: Stem/Stromal Cellular Isolation (Digestive); Procedure: HD-PRP (High Density Platelet Rich Plasma); Procedure: Emulsified AD-tSVF; Procedure: Emulsified AD-cSVF

INTERVENTIONS:
Procedure: Intradermal Injection in hair loss — Comparative Injection of Control (PRP & Acel) in hair loss; 2) Intradermal Injection in hair loss
  Other Names: ARM 1; Matricell (ACell); Platelet Rich Plasma
Procedure: Platelet Rich Plasma — Growth factors and cytokines to promote healing and vascular supply
  Other Names: ARM 1, ARM 2, ARM 3
Procedure: Adipose Derived Stem/Stromal Cells — Harvesting Adipose Lipoaspirate with Microcannula System
  Other Names: ARM 2 and ARM 3; Platelet Rich Plasma; Emulsification of Adipose Derived tSVF; Intradermal Injection in hair loss
  Arms: ARM 2; ARM 3
Procedure: Stem/Stromal Cellular Isolation (Digestive) — Cell isolation and concentration add back to AD-stem/stromal cells utilizing Centricyte 1000 Protocol
  Other Names: ARM 3; Platelet Rich Plasma; Emulsification of Adipose Derived cSVF; Intradermal injection in hair loss
  Arms: ARM 3
Procedure: MatriStem Matrix (ACell) - Current Standard of Care
  Arms: ARM 1
Procedure: HD-PRP (High Density Platelet Rich Plasma)
Procedure: Emulsified AD-tSVF
  Arms: ARM 2; ARM 3
Procedure: Emulsified AD-cSVF — Stem/Stromal Cellular Isolate Added Back to Emulsified AD-tSVF
  Arms: ARM 3

SUMMARY:
Purpose The primary objective of this study is to evaluate the safety and efficacy of the use of a biocellular mixture of emulsified adipose-derived tissue stromal vascular fraction (AD-tSVF) and high density platelet-rich plasma concentrate (HD- PRP) as compared with adipose-derived cell-enriched SVF (AD-cSVF) + AD-tSVF and HD- PRP concentrates in treatment of androgenetic alopecia (AGA) and Female Pattern Hair Loss (FPHL).

Assigned Interventions

1. HD-PRP + Matristem Matrix (ACell)
2. Experimental: HD-PRP + Emulsified AD-tSVF
3. Experimental: HD- PRP + Emulsified AD-tSVF + Emulsified AD-cSVF Device: Tulip Microcannula Closed Syringe For All Lipoaspiration (2.11 mm Diameter, offset Carraway) Centrifugation technique to acquire concentrated platelets (per manufacturer's approved protocol) Healeon ACM Emulsification System that prepares microcannula harvested AD-tSVF for small needle (25g) retrograde threaded intradermal scalp injection.

Healeon Centricyte 1000 system for cellular isolation of AD-cSVF from AD-tSVF and testing by Flow Cytometry (ORFLO MoxiFlow) Procedure: Closed syringe microcannula lipoaspiration (AD-tSVF) Procedure: Emulsification of AD-tSVF via Healeon ACM Protocol (Newbury Park, CA, USA) Procedure: Biocellular mix of emulsified AD-tSVF and HD-PRP for intradermal injection in scalp; (Arm 2) Procedure: Cellular isolation (AD-cSVF) Centricyte 1000 incubation/shaker system using GMP certified, sterile Liberase MNP-S (Roche #06297790001) for enzymatic digestion manufacturer standard protocol. Creation of emulsified AD-tSVF + PRP + cell-enriched AD-cSVF for intradermal injection in scalp (Arm 3) Sham Comparator: No Fat Control using Emcyte II PRP Concentrate + Matristem (Acell) for subcutaneous scalp injection patterned per square centimeter of scalp. Procedure: Emcyte Pure PRP® II system to concentrate Platelets via using manufacturer standard protocol

DETAILED DESCRIPTION:
Detailed Description:

The cosmetic discipline of hair restoration is rooted in numerous landmark studies and progressive medical science in the medical literature. , , , , With the advent of advance theories and science within the scope of regenerative medicine, numerous reports are noted in the literature. , , , , , using biological modalities, e.g., HD-PRP concentrates defined as > 4-6 times patient circulating baselines, for stimulation of scalp tissues and hair follicles in androgenetic alopecic (AGA).

Design of this study is intended to be a prospective, randomized, multicenter trial with blinding of outcomes for independent observer, clinical provider and patient observation/satisfaction studies. The study proposes adipose-derived (AD) biocellular material when mixed with platelet high density concentrates (HD-PRP) offers a potential advantage for a markedly more effective therapeutic profile in areas of follicular miniaturization, tissue age related senescence, and effect the decreased vascular capabilities by stimulation of vasculoneogenesis. The benefits of using autologous adipose-derived stem/stromal cell (ADSCs) populations are cell proliferation and vasculogenesis that is intrinsically linked with native immunomodulatory capacities. Reports describing the safety and efficacy of this biocellular combination have been reported in peer reviewed literature. , In the second and third arm of this study, the use of regenerative protocols currently being utilized in the treatment of degenerative musculoskeletal conditions is employed. These protocols feature the use of an emulsified AD-tSVF and emulsified cell enriched AD-cSVF containing the full heterogeneous stem/stromal cell population and matrix that is injected into the regions of scalp containing the microenvironment (niche) of the hair follicle. In Arm 3, cellular enrichment of the emulsified AD-tSVF is accomplished via a semi-automated, closed sterile system (Healeon CentriCyte 1000 system) to isolate and concentrate AD-cSVF. The AD-cSVF is then mixed with high-density platelet rich plasma (HD-PRP) concentrates and emulsified AD-tSVF tissues (AD-tSVF) prior to scalp injection. This injected cell-enriched product contains native adipose tissue scaffolding, autologous HD-PRP, and enriched adipose stem/stromal cell-enriched concentration of stromal/stem cells (AD-cSVF).

The goal of this study is to demonstrate the safety and efficacy of the HD-PRP + AD-tSVF + AD-cSVF biocellular injections into the scalp of men and women with a diagnosis of non-scaring alopecias, with full reporting of AE and SAE (adverse events). The biocellular material is injected 3-5 mm in depth within the mid-reticular dermis to upper subcutaneous fat layer of the scalp for the purpose of regenerating the miniaturized hair follicle, and delivering a milieu of stromal/stem cells that facilitate regenerative changes within the tissue sites. In addition to providing tissue scaffolding, and a greater number of stromal/stem cells to the tissues surrounding the follicular niche, the novel use and emulsification of AD tissues with cell-enriched biocellular material permits ergonomic facilitation of layered injection patterns in the scalp with small gauge (25-27 gauge) needles This emulsified AD Biocellular methodology reduces injection pressure requirements using smaller gauge needles. When clinically compared to the use of much larger needles required to inject non-emulsified AD-tSVF, it is an improvement on current techniques.

Successful stem/stromal cell-enrichment of AD-tSVF and HD PRP biocellular mixture has been reported in numerous peer-reviewed and published clinical experiences of injections for structural tissue augmentation in plastic surgery, chronic wound therapies, and ultrasound guided musculoskeletal treatments in orthopedic surgery. A "retrograde" filling technique creating a potential space and subsequently injecting into this space the biocellular material as the needle is withdrawn is advanced in this study.

All patients will undergo venipuncture for obtaining HD-PRP concentrates following FDA approved Emcyte II manufacturer's guidelines. Those patients having biocellular treatment with also undergo a small volume closed syringe microcannula lipoaspiration to acquire AD-tSVF tissues, which will be emulsified via the Healeon ACM System per manufacturer's guidelines. Cellular testing of samples in Arm 2 and Arm 3 will be performed by flow cytometry (ORFLO, MoxiFlow, Ketchum, ID, USA) for viability and cell concentrations. The trial will include the biocellular mixture of HD-PRP + emulsified AD-tSVF (Arm 2) and/or, HD-PRP + emulsified AD-tSVF + AD-cSVF (Arm 3). Study will utilize a standardized high-density PRP concentration system on all patients in the same volume. The definition of HD-PRP concentrates is a minimum =/>4 times patient circulating platelet counts.

A detailed patient medical history, informed consent, and screening evaluation will determine eligibility and candidacy for the study. Each patient will undergo a small volume lipoaspiration (defined as <100 cc) under local anesthesia with, or without, oral sedation. Candidates will be assigned to one of three treatment ARMs. The treatment ARMS are: ARM 1: HD-PRP + Matristem Matrix (A-Cell) (control); ARM 2: HD-PRP + emulsified AD-tSVF; and, ARM 3: HD-PRP + emulsified AD-tSVF + cell-enriched AD-cSVF. All patients will receive a standard ring block local anesthesia of the scalp treatment areas, followed by retrograde injection pattern of the biocellular material.

Recording of the platelet baseline and treatment concentrates, flow cytometric examination of cell viability, and cell counts of AD-cSVF will be completed on each patient. Biocellular injections and treatment will be given on two (2) separate procedures three (3) months apart. Follow up clinical examinations are to be performed at 6 months and 1year period with completion of outcomes analyses including independent observer, clinician, and subject satisfaction. The volume of the HD-PRP concentrates will be the standardized in volume for all trial ARMs.

Immediate reporting to the study group for all AR and SAR will be documented and recorded for the safety records directly to Ken Williams, DO, as Principal Clinical Investigator. This Clinical Trial will have a sample size of 60 patients at up to six (6) centers utilizing the same protocols, equipment and reporting requirements.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Males with a diagnosis of Androgenetic Alopecia (AGA).
  2. Females with a biopsy proven diagnosis of Female Pattern Hair Loss (FPHL) excluding scaring or autoimmune disorders.
  3. Males with hair loss consistent with Grades II, III, IIIA, III-Vertex, IV, IV-A, based on Norwood-Hamilton Scale.
  4. Females with hair loss consistent with Grades I-3, I-4, II-1, II-2 based on the Savin Scale.
  5. Demonstrated ability to legally provide written informed consent and comply with the study requirements
  6. For women of childbearing potential with screening negative pregnancy test and subject agrees to avoid pregnancy with two forms of contraception for the duration of study
  7. Subject is willing to maintain existing and consistent hair length and color.
  8. Ability to complete study procedures, patient surveys, and photodocumentation.
  9. Subject is ≥ 18 years of age.
  10. Five (5) year cancer free period without treatment and no evidence of recurrence

Exclusion Criteria:

1. Subjects who have used oral spironolactone, finasteride, dutasteride, minoxidil, or any oral or topical medication including over the counter and herbal medications for the treatment of hair loss within 12 months of study screening.
2. Simultaneous treatment with an investigational product or procedure within 30 days, or planned future participation in another clinical study
3. Subject has previously failed or has been deemed non-responsive to a previous experimental hair loss treatment.
4. Subject must have no previous hair transplant, PRP, biocellular treatments, micro needling, cold laser therapies, or any other scalp or hair loss treatment.
5. Subject with previously diagnosed or suspected of having active scaring alopecia, autoimmune diseases such as serum lupus erythematosus, or alopecia areata; unspecified dermatologic condition, or disorders that will make hair growth difficult (such as systemic burns, etc.).
6. History of or active diagnosis of autoimmune disease or organ transplantation or immunosuppressive medication(s).
7. Receiving active cancer treatment or have present or previous malignancies except a history of squamous or basal skin cell carcinoma with excision for cure.
8. Active systemic infection at the time of enrollment. If acquired afterwards, exclusion based on clinical judgment of investigator.
9. Use of chronic antibiotics and/or systemic corticosteroids.
10. Use of systemic agents that increase bleeding or clotting, or disorders associated with these effects, including patients receiving GIIB/IIIa inhibitors in the 2 weeks prior to the study procedure through to 1 week after the study procedure.
11. Clinically significant or current medical or psychiatric illness.
12. Prior surgery in the treatment area.
13. Any disease or condition (medical or surgical) that, in the opinion of the investigator, might compromise dermatologic, hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system function; or any condition that would place the subject at increased risk of increased morbidity or mortality.
14. Pregnant or lactating female, or women trying to become pregnant.
15. Known allergic reaction to components of study treatment and/or study injection procedure
16. Subject has any disorder or any reason that may prevent compliance to study procedures and visits.
17. Employees or family members of the study staff.
18. Untreated or uncontrolled thyroid disorder (abnormal TSH/free T4) or diabetes mellitus (HgbA1C > 8.0).
19. Subject who has a sensitive, irritated, or abraded scalp area.
20. Women who have an alternate diagnosis that is associated with hair loss.
21. Clinically significant abnormal findings on laboratory screening panels:

    * Hemoglobin ≤ 10 g/dL
    * Hepatic dysfunction, as defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin levels > 1.5 times the upper limit of normal range prior to randomization.
    * Chronic renal insufficiency as defined as a serum creatinine > 1.2 mg/dL for women and > 1.5 mg/dL for men.
    * An elevated PT/PTT, INR,
    * platelet count < 100 x 109/L

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-14 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety-Tolerability Assess of SAE/AE Assessment of SAE/AES | 6 months
  Safety-Tolerability Assess of SAE/AE

SECONDARY OUTCOMES:
Hair Growth Trichogram | 12 Months
  Growth Assessment by Trichogram [ Designated as safety issue: No ] Assessment by Trichogram
Hair Density Trichogram | 12 Months
  Hair Density Assessment Trichogram [ Designated as safety issue: No ] Assessment by Trichogram
Global Photometric Scalp Hair | 12 Months
  Global Photographic assessment scalp hair Photographic assessment of scalp hair by independent observer
Hair Investigator Satisfaction | 12 Months
  Hair Investigator Satisfaction Survey [ Designated as safety issue: No ] Assessment of treatment outcome by treating physician
Patient Satisfaction Survey | 12 Months
  Patient Satisfaction Survey [Designated as safety issue: No] Assessment of treatment Outcomes by patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Welter, MD, PhD, MD,PhD, Study Director — Regeneris; Marco Barusco, MD, Study Director — Brusco Clinic; Kenneth Williams, DO, Principal Investigator — Irvine Institute Medicine & Cosmetic Surgery
Locations (1):
- Kenneth Williams, DO, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Understanding Adipose-derived Stromal Vascular Fraction (AD-SVF) Cell Biology and Use on the Basis of Cellular, Chemical, Structural and Paracrine Components: A Concise Review
- [Background] Alexander RW, Harrell DB. Autologous fat grafting: use of closed syringe microcannula system for enhanced autologous structural grafting. Clin Cosmet Investig Dermatol. 2013 Apr 8;6:91-102. doi: 10.2147/CCID.S40575. Print 2013. PMID 23630430
- [Background] Understanding Mechanical Emulsification (Nanofat) Versus Enzymatic Isolation of Tissue Stromal Vascular Fraction (tSVF) Cells from Adipose Tissue: Potential Uses in Biocellular Regenerative Medicine
- [Background] Zuk, P., Adipose-Derived Stem Cells in Tissue Regeneration. Review, Hindawi Publlishing Coripration, ISRN Stem Cells, Volume 2013, Artilce ID 713959, http://dx.doi.org/10.1155/2013/713959
- [Background] Tobita M, Tajima S, Mizuno H. Adipose tissue-derived mesenchymal stem cells and platelet-rich plasma: stem cell transplantation methods that enhance stemness. Stem Cell Res Ther. 2015 Nov 5;6:215. doi: 10.1186/s13287-015-0217-8. PMID 26541973